CLINICAL TRIAL: NCT02540031
Title: The Impact of Additional Oral Preparation on the Quality of Bowel Preparation for Colonoscopy in Patients Showing Brown Effluents
Brief Title: The Impact of Additional Oral Preparation on the Quality of Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-06-014-003
Record Dates: First submitted 2015-08-08; First posted 2015-09-03 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Bowel Preparation Quality

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Additional oral preparation (Experimental): The investigational or experimental arm will receive standard oral preparation plus additional oral preparation (1l of polyethylene glycol (PEG)+ascorbic acid (Asc)) for colonoscopy.
  * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  Interventions: Drug: Additional oral preparation (3L of PEG+Asc, "Coolprep®")
- Standard oral preparation (Active Comparator): The control arm will receive currently used oral preparation (2L of polyethylene glycol+ascorbic acid) for colonoscopy.
  * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  Interventions: Drug: Standard oral preparation (2L of PEG+Asc, "Coolprep®")

INTERVENTIONS:
Drug: Additional oral preparation (3L of PEG+Asc, "Coolprep®") — The interventional or experimental arm will receive 1l of additional PEG+Asc, "Coolprep®" on the day of colonoscopy
  * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  Other Names: Coolprep® (TaeJoon Pharmaceuticals, Seoul, Korea):3L
  Arms: Additional oral preparation
Drug: Standard oral preparation (2L of PEG+Asc, "Coolprep®") — The control arm will receive currently used oral preparation (2l of PEG+Asc, "Coolprep®") for colonoscopy
  * Compositions/1L : Sodium Chloride 2.691g Potassium Chloride 1.015g Anhydrous sodium sulfate 7.5g PEG 3350 100g ascorbic acid 4.7g sodium ascorbate 5.9g
  Other Names: Coolprep® (TaeJoon Pharmaceuticals, Seoul, Korea) : 2L
  Arms: Standard oral preparation

SUMMARY:
Although adequate bowel preparation is essential for successful colonoscopy, the 23% of patients had shown inadequate bowel preparation. Inadequate bowel preparation may results in incomplete examination, increased patient's discomfort, decreased polyp detection rates, ultimately leading to repeated colonoscopies. One prior study showed that patients reporting their last rectal effluents as brown color or solid stool had a 54% chance of having fair or poor preparation. Thus, recent consensus guideline suggested consideration of additional oral preparation in patients presenting brown effluents on the day of colonoscopy. However, the data supporting additional oral preparation is still spares. Therefore, the investigators aimed to examine the impact of additional oral preparation on the quality of bowel preparation for colonoscopy in patients showing brown effluents on the day of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients who reporting their last rectal effluents as brown color or solid stool on the day colonoscopy

Exclusion Criteria:

* known hypersensitivity to polyethylene glycol
* severe congestive heart failure [New York Heart Association (NYHA) grade III or grade IV]
* severe renal insufficiency (creatinine clearance <30 ml/min)
* hemodynamic instability
* suspected intestinal obstruction or perforation
* compromised swallowing reflex or altered mental status
* pregnancy or lactating woman
* patients who declined to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | Day 1
  The primary outcome will be the endoscopist's assessment of the quality of preparation using a standardized bowel preparation scale

SECONDARY OUTCOMES:
Adenoma detection rate | Day 1
  Number of adenomatous polyps
Patient compliance | Baseline
  Patient compliance with preparation instructions self-reported in a pre-procedure questionnaire
Patient satisfaction | Baseline
  Patient's perception of the preparation method as self-reported on a pre-procedure questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

REFERENCES:
- [Result] Fatima H, Johnson CS, Rex DK. Patients' description of rectal effluent and quality of bowel preparation at colonoscopy. Gastrointest Endosc. 2010 Jun;71(7):1244-1252.e2. doi: 10.1016/j.gie.2009.11.053. Epub 2010 Apr 1. PMID 20362286